CLINICAL TRIAL: NCT03382353
Title: Efficacy of Multiple Nonpharmacological Interventions in Individuals With Subjective Memory Complaints
Brief Title: EMuNI Project: Multiple Nonpharmacological Interventions
Acronym: EMuNI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Centro San Giovanni di Dio Fatebenefratelli (Other)
Collaborators: Ospedale San Raffaele (Other); Istituto Di Ricerche Farmacologiche Mario Negri (Other)
Responsible Party: Principal Investigator, Enrica Cavedo, Principal Investigator, IRCCS Centro San Giovanni di Dio Fatebenefratelli
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GR-2011-02350494
Record Dates: First submitted 2017-12-09; First posted 2017-12-22 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Lifestyle Risk Reduction
Keywords: primary prevention; Subjective Cognitive Decline; Neuroimaging; Alzheimer's disease; nonpharmacological interventions; multidomain lifestyle interventions
MeSH Terms: conditions — Risk Reduction Behavior; Alzheimer Disease | interventions — Dietary Supplements; Training Support; Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No Treatment (NT) (Active Comparator): Educational training
  Interventions: Behavioral: Educational training
- Partial Treatment (PT) (Experimental): Nutritional supplementation & Counselling on a brain-healthy diet
  Interventions: Dietary Supplement: Nutritional supplementation; Behavioral: Counselling on a brain-healthy diet
- Full Treatment (FT) (Experimental): Nutritional supplementation & Counselling on a brain-healthy diet & Physical exercise training & Computerized cognitive training
  Interventions: Dietary Supplement: Nutritional supplementation; Behavioral: Counselling on a brain-healthy diet; Behavioral: Physical exercise training; Behavioral: Computerized cognitive training

INTERVENTIONS:
Dietary Supplement: Nutritional supplementation — Daily consumption of Tramiprosate (100 mg) for 1 year
  Arms: Full Treatment (FT); Partial Treatment (PT)
Behavioral: Educational training — 16 educational lessons (twice a week): basic principles of different cognitive domains (e.g. memory, attention, perception) and educational DVD viewing.
  Arms: No Treatment (NT)
Behavioral: Counselling on a brain-healthy diet — 4 lessons on the principles of Mediterranean Diet lead by a nutritionist, aimed to teach how to include brain-healthy foods in daily diet (e.g. antioxidant, omega-3 fatty acids and vitamins). Each participant will receive the educational material presented.
  Arms: Full Treatment (FT); Partial Treatment (PT)
Behavioral: Physical exercise training — 80 sessions of physical exercise supervised by a Fitness Training Expert with the aim of achieving 150 minutes of moderate-intensity physical activity per week
  Arms: Full Treatment (FT)
Behavioral: Computerized cognitive training — 16 cognitive training sessions (twice a week) supervised by a psychologist, aimed to improve Attention, Processing speed, Memory, Social skills and Intelligence using BrainHQ (www.brainhq.com).
  Arms: Full Treatment (FT)

SUMMARY:
By 2030, the global prevalence of Alzheimer's Disease (AD) is predicted to reach 65.7 million worldwide. Despite extensive research efforts, a cure for AD has not been identified. Recent studies on non-demented individuals have demonstrated the importance of a healthy lifestyle (physical exercise, healthy diet) and non pharmacological interventions (diet supplements) to delay the onset of the cognitive decline (Vemuri P et al., 2012). Given that AD is a multi-factorial disorder, some multi- component interventions at early stages could be the best strategy currently available to delay the AD onset. The aim of this study is to investigate the effects of combined non-pharmacological interventions, at different levels of intensity, on cognitive performance, on basic (hippocampal, brain ventricle volumes and white matter lesions) and advanced magnetic resonance imaging (MRI) markers (Resting-state Functional MRI, Probabilistic Diffusion Tensor Tractography

DETAILED DESCRIPTION:
BACKGROUND Recent evidence showed that aerobic exercise, dietary habits and nutritional supplements consumption seem essential for maintaining good cognitive performances increasing hippocampal volume (HV) in healthy elderly people (Erickson et al., 2011; Bowman et al., 2012). Computerized cognitive trainings are effective in improving cognitive functions of healthy older adults (Lampit et al., 2014). Subjective memory complaint (SMC) individuals showed HV, white matter lesions (WML) and brain ventricle volumes (BVV) at limits of normative population (Cavedo et al., 2012) supporting the hypothesis that they are persons at risk of AD (Sperling et al., 2011). The above non-pharmacological treatments, when separately applied, do not impact on cognition and neuropathological processes of AD. On the contrary, combined treatments, in persons at risk to develop AD, could represent the first line of intervention to delay the onset of cognitive impairment.

SPECIFIC AIMS

1. To investigate the combined effect of aerobic exercise, dietary habits, nutritional supplements, and cognitive training administered at three different levels of intensity on cognitive performance in subjective memory complaints individuals. The three different intensity levels of nonpharmacological treatments will be organized as follows: (i) No Treatment (NT) will include educational training (sham condition); (ii) Partial Treatment (PT) will include exclusively the consumption of a nutritional supplement and a training for a balanced diet; (iii) Full treatment (FT) will include all above condition plus computerized cognitive training (no sham condition) and aerobic fitness training.
2. To investigate the effect of the above treatments (NT, PT, FT) on basic markers of magnetic resonance imaging (MRI) such as HV, WML and Brain Ventricle Volume (BVV) in subjective memory complaints individuals.
3. To investigate the effect of NT, PT and FT on advanced MRI markers such as structural brain connectivity and brain resting networks in subjective memory complaints individuals.

HYPHOTESIS AND SIGNIFICANCE An improvement in cognitive performances, basic (HV, WML, BVV) and advanced (structural brain connectivity and brain resting networks) MRI markers will be expected in FT group compared to NT group. Moreover, the investigators hypothesize an effect dependent of the number of combined treatments, thus the PT group is expected to show intermediate results (among NT and FT groups) in the cognitive performances, basic and advanced MRI markers previously described.

ELIGIBILITY:
Inclusion Criteria:

* age between 60 and 80 years;
* presence of memory complaints

Exclusion Criteria:

* objective cognitive impairment on standard neuropsychological testing;
* history of psychiatric disorders or current clinically relevant depressive or anxious symptoms;
* pacemakers, cochlear implant, metal inserts in the head or shoulders

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-01; Primary Completion 2017-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Cognitive functions | 12 months
  Neuropsychological test performances

SECONDARY OUTCOMES:
Basic imaging marker 1 | 12 months
  Hippocampal volumes
Basic imaging marker 2 | 12 months
  White matter hyperintensities volumes
Basic imaging marker 3 | 12 months
  Brain ventricle volumes

OTHER OUTCOMES:
Advanced imaging marker 1 | 12 months
  Structural brain connectivity
Advanced imaging marker 2 | 12 months
  Functional networks connectivity at rest

CONTACTS AND LOCATIONS:
Overall Officials: Enrica Cavedo, PhD, Principal Investigator — IRCCS Centro San Giovanni di Dio Fatebenefratelli
Locations (2):
- Italy (2):
  - IRCCS Centro San Giovanni di Dio Fatebenefratelli, Brescia
  - Ospedale San Raffaele, Milan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bowman GL, Silbert LC, Howieson D, Dodge HH, Traber MG, Frei B, Kaye JA, Shannon J, Quinn JF. Nutrient biomarker patterns, cognitive function, and MRI measures of brain aging. Neurology. 2012 Jan 24;78(4):241-9. doi: 10.1212/WNL.0b013e3182436598. Epub 2011 Dec 28. PMID 22205763
- [Background] Cavedo E, Galluzzi S, Pievani M, Boccardi M, Frisoni GB. Norms for imaging markers of brain reserve. J Alzheimers Dis. 2012;31(3):623-33. doi: 10.3233/JAD-2012-111817. PMID 22672878
- [Background] Erickson KI, Voss MW, Prakash RS, Basak C, Szabo A, Chaddock L, Kim JS, Heo S, Alves H, White SM, Wojcicki TR, Mailey E, Vieira VJ, Martin SA, Pence BD, Woods JA, McAuley E, Kramer AF. Exercise training increases size of hippocampus and improves memory. Proc Natl Acad Sci U S A. 2011 Feb 15;108(7):3017-22. doi: 10.1073/pnas.1015950108. Epub 2011 Jan 31. PMID 21282661
- [Background] Lampit A, Hallock H, Valenzuela M. Computerized cognitive training in cognitively healthy older adults: a systematic review and meta-analysis of effect modifiers. PLoS Med. 2014 Nov 18;11(11):e1001756. doi: 10.1371/journal.pmed.1001756. eCollection 2014 Nov. PMID 25405755
- [Background] Sperling RA, Aisen PS, Beckett LA, Bennett DA, Craft S, Fagan AM, Iwatsubo T, Jack CR Jr, Kaye J, Montine TJ, Park DC, Reiman EM, Rowe CC, Siemers E, Stern Y, Yaffe K, Carrillo MC, Thies B, Morrison-Bogorad M, Wagster MV, Phelps CH. Toward defining the preclinical stages of Alzheimer's disease: recommendations from the National Institute on Aging-Alzheimer's Association workgroups on diagnostic guidelines for Alzheimer's disease. Alzheimers Dement. 2011 May;7(3):280-92. doi: 10.1016/j.jalz.2011.03.003. Epub 2011 Apr 21. PMID 21514248
- [Background] Vemuri P, Lesnick TG, Przybelski SA, Knopman DS, Roberts RO, Lowe VJ, Kantarci K, Senjem ML, Gunter JL, Boeve BF, Petersen RC, Jack CR Jr. Effect of lifestyle activities on Alzheimer disease biomarkers and cognition. Ann Neurol. 2012 Nov;72(5):730-8. doi: 10.1002/ana.23665. PMID 23280791
- [Derived] Rolandi E, Dodich A, Mandelli S, Canessa N, Ferrari C, Ribaldi F, Munaretto G, Ambrosi C, Gasparotti R, Violi D, Iannaccone S, Marcone A, Falini A, Frisoni GB, Galluzzi S, Cerami C, Cavedo E. Targeting brain health in subjective cognitive decline: insights from a multidomain randomized controlled trial. Aging Clin Exp Res. 2025 May 14;37(1):151. doi: 10.1007/s40520-025-03062-z. PMID 40366507